CLINICAL TRIAL: NCT03031912
Title: A Phase 2 Randomized, Multi-Center Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine Candidate in HIV-Infected Adults and Adolescents
Brief Title: African-Canadian Study of HIV-Infected Adults and a Vaccine for Ebola - ACHIV-Ebola
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry); International Development Research Centre, Canada (Other Government); Dalhousie University (Other); Université de Montréal (Other); Coalition for Epidemic Preparedness Innovations (Other); University of Ottawa (Other); Centre Muraz (Other); Institute for Health Research - Epidemiological Surveillance and Training (IRESSEF) (Unknown)
Responsible Party: Principal Investigator, Joanne Langley, COORDINATING Investigator, Canadian Immunization Research Network
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CT1401-B
Record Dates: First submitted 2016-12-22; First posted 2017-01-26 (Estimated); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Ebola
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Ebola Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: V920 (Active Comparator): Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  Interventions: Biological: V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine
- Group 2: Placebo (Placebo Comparator): Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Interventions: Other: Saline

INTERVENTIONS:
Biological: V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine — The rVSVΔG-ZEBOV-GP vaccine is a live attenuated recombinant virus consisting of a single recombinant VSV isolate (11481 nt, strain Indiana) with the gene for the Zaire ebolavirus GP (ZEBOV GP), Kikwit strain replacing the gene for the VSV GP, which has been deleted. This results in a VSV backbone with the ZEBOV GP constituting the envelope of the virus.
  Arms: Group 1: V920
Other: Saline — Normal saline (0.9%) has been chosen as an inert substance to serve as placebo control.
  Arms: Group 2: Placebo

SUMMARY:
This is a randomized, placebo-controlled, multi-site, double-blind trial of V920 (rVSVΔG-ZEBOV-GP) Ebola Virus vaccine candidate in subjects with HIV infection to be conducted in conformance with Good Clinical Practices. The study will take place at 2 Canadian sites (Centre Hospitalier de l'Université de Montréal and Ottawa General Hospital) and 2 African sites (Centre MURAZ, Burkina Faso and Centre Hospitalier National Aristide Le Dantec, Dakar, Senegal). The Duration of Study: 365 days for each participant not including screening.

DETAILED DESCRIPTION:
The study will enroll approximately 250 participants, ~100 at 2 sites in Canada and ~100 at 2 sites in Africa. Overall ~200 participants will receive the study vaccine and 50 will receive a placebo . Sequential enrollment of five study cohorts will occur over time at each study site according to CD4 T-cell counts: Group 1 will include adult subjects with CD4 ≥ 500 cells/mm3, Group 2 CD4 > 350 and < 500 cells/mm3, Group 3 CD4 ≥ 200 and ≤ 350 cells/mm3, Group 4 adolescents CD4 ≥ 200 cells/mm3, and Group 5 adults and adolescents CD4 ≥ 200 cells/mm3. Enrolment and vaccine administration will begin with the group with the highest CD4 count. When the D42 post-vaccination period is completed for all subjects in Group 1, and the Data Safety Monitoring Board (DSMB) has reviewed the safety data and determined that there are no concerns, enrolment and vaccination of the next CD4 cohort may begin. Similarly, when the D42 safety data for Group 2 has been reviewed/approved by the DSMB, enrolment and vaccination of participants in Group 3 may begin. Adolescents 13-17 years of age (inclusive) with CD4 ≥ 200 will be enrolled after D42 safety is reviewed in adults with CD4 ≥ 200. Adolescents 13-17 years of age (inclusive) and adults with CD4 ≥ 200 will be enrolled after D42 safety is reviewed in adolescents with CD4 ≥ 200.Within each group, participants will be randomly assigned to receive one dose of ≥2 x 107 pfu of the study vaccine or the placebo in a ratio of 4 to 1 (160:40). Participants will complete memory aids for 42 days following vaccination.

Specific procedures to be performed during the trial, as well as their prescribed times and associated visit windows, are outlined in the Trial Flow Chart - Section 6.0. Details of each procedure are provided in Section 7.0 - Trial Procedures.

This trial will use an adaptive design based on pre-specified criteria, using an independent, external DSMB to monitor safety and immunogenicity. There will be 3 formal safety analyses performed by the DSMB. Data for at least 75% of participants must be available for each analysis. The first safety analysis will be conducted when the first group (CD4 ≥ 500 cells/mm3) will have completed 42 days of follow-up post vaccination. The second safety analysis will be conducted when the second group (CD4 > 350 and < 500 cells/mm3) will have completed 42 days of follow-up post vaccination. The third safety analysis will be conducted when the third group (Adults CD4 ≥ 200 and ≤ 350 cells/mm3) will have completed 42 days of follow-up post vaccination. The fourth safety analysis will be conducted when the fourth group (Adolescents CD4 ≥ 200) will have completed 42 days of follow-up post vaccination.

Results of the safety analysis will be reviewed by the DSMB, which will make recommendations to the Sponsor to continue, modify or end the trial according to the plan described briefly in Section 2.2 - Trial Diagram and in detail in Section 8.0 - Statistical Analysis Plan. In case of an outbreak of Ebola Zaire the DSMB may recommend to vaccinate subjects randomized to receive placebo with V920 provided at least 84 days of SAE follow-up is conducted.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adult or adolescent male or non-pregnant, non-breastfeeding female, ages 13 to 65 (inclusive) at the time of screening;
* On antiretroviral therapy with an undetectable viral load (< 40 c/ml);
* CD4 T cell counts ≥ 200 cells/mm3;
* Written informed consent (subject or parent) and assent (adolescent), after reading the consent form and having adequate opportunity to discuss the study with an investigator or a qualified designee
* Free of clinically significant health problems that could affect the safety of the participant, as determined by the Investigator by pertinent medical history and clinical examination prior to entry into the study;
* Available, able, and willing to participate for all study visits and procedures;
* Males and females who are willing to practice abstinence from sexual intercourse, or are willing to use effective methods of contraception, from at least 30 days prior to vaccination until 2 months after vaccination.

  1. If the female partner is NOT of childbearing potential, the couple will only be required to use condoms, without other adjunctive contraception.
  2. For this study, a woman is considered of childbearing potential unless postmenopausal (≥ 1 year without menses) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy)
  3. Effective contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label for example:

  i. Male condoms PLUS: ii. Oral contraceptives, either combined or progestogen alone iii. injectable progestogen iv. implants of etenogestrel or levonorgestrel v. oestrogenic vaginal ring vi. percutaneous contraceptive patches vii. intrauterine device or intrauterine system
* Be willing to minimize blood and body fluid exposure of others for 6 weeks after vaccination

  1. Use of effective barrier prophylaxis, such as latex condoms, during penetrative sexual intercourse
  2. Avoiding the sharing of needles, razors, or toothbrushes
  3. Avoiding open-mouth kissing

Exclusion Criteria:

* History of prior infection with a filovirus or prior participation in a filovirus vaccine trial;
* History of prior infection with VSV or receipt of a VSV-vectored vaccine;
* Is a healthcare worker who has direct contact with patients
* Presence of any febrile illness or any known or suspected acute illness on the day of any first immunization (subject may be rescheduled);
* Clinical manifestations of systemic diseases considered by the investigator to impact safety or immunogenicity
* Receipt of systemic glucocorticoids (a dose ≥ 20 mg/day prednisone or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within six months;
* Receipt of any investigational drug within 12 months of vaccination;
* Receipt of any live virus vaccine within 42 days prior to study entry or any other (non-live virus) vaccine within 14 days prior to study entry.
* History of sensitivity to any component of study vaccines per investigator brochure or package insert;
* Any baseline laboratory screening tests which is outside of acceptable range as defined in the protocol: ALT, AST, creatinine, hemoglobin, platelet count, total white blood cell count, urine protein, urine occult blood, urine glucose (Appendix 2). To exclude transient abnormalities, the investigator may repeat a test up to twice, and if the repeat test is normal, subject may be enrolled;
* Have an active malignancy or history of metastatic or hematologic malignancy except non-melanoma skin cancers;
* Suspected or known alcohol and/or illicit drug abuse within the past 5 years;
* Moderate or severe illness and/or fever >101°F (38.3ºC) within one week prior to vaccination;
* Pregnant or breastfeeding female, or female who intends to become pregnant during the study period;
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period;
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Tremblay, MD, Principal Investigator — CHUM
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Changes made as requested by PRS team. Results have been provided for each arm of each cohort.
Groups:
- Cohort 1: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  ≥500 cells/mm3
  Adults.
- Cohort 1: Placebo: Participants randomly assigned to receive placebo control.
  ≥500 cells/mm3
  Adults.
- Cohort 2: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  >350 and <500 cells/mm3
  Adults.
- Cohort 2: Placebo: Participants randomly assigned to receive placebo control.
  >350 and <500 cells/mm3
  Adults.
- Cohort 3: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  ≥200 and ≤350 cells/mm3
  Adults.
- Cohort 3: Placebo: Participants randomly assigned to receive placebo control.
  ≥200 and ≤350 cells/mm3
  Adults.
- Cohort 4: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  ≥200 cells/mm3
  Adolescents.
- Cohort 4: Placebo: Participants randomly assigned to receive placebo control.
  ≥200 cells/mm3
  Adolescents.
- Cohort 5: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  ≥200 cells/mm3
  Adults and adolescents.
- Cohort 5: Placebo: Participants randomly assigned to receive placebo control.
  ≥200 cells/mm3
  Adults and adolescents.
Period: Overall Study
Arm/Group | Cohort 1: V920 | Cohort 1: Placebo | Cohort 2: V920 | Cohort 2: Placebo | Cohort 3: V920 | Cohort 3: Placebo | Cohort 4: V920 | Cohort 4: Placebo | Cohort 5: V920 | Cohort 5: Placebo
Started | 41 | 10 | 40 | 10 | 41 | 9 | 40 | 10 | 40 | 10
Completed | 40 | 9 | 40 | 9 | 41 | 9 | 40 | 10 | 40 | 10
Not Completed | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine
  Adults: CD4 cells/mm3 ≥ 500
  1
- Cohort 1: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adults: CD4 cells/mm3 ≥ 500
  1
- Cohort 2: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine
  Adults: CD4 cells/mm3 >350 and < 500
- Cohort 2: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adults: CD4 cells/mm3 >350 and < 500
- Cohort 3: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine
  Adults: CD4 cells/mm3 ≥ 200 and ≤ 350
- Cohort 3: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adults: CD4 cells/mm3 ≥ 200 and ≤ 350
- Cohort 4: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine
  Adolescents: CD4 cells/mm3 ≥ 200
- Cohort 4: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adolescents: CD4 cells/mm3 ≥ 200
- Cohort 5: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine
  Adults and adolescents: CD4 cells/mm3 ≥ 200
- Cohort 5: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adults and adolescents: CD4 cells/mm3 ≥ 200
- Total: Total of all reporting groups
Arm/Group | Cohort 1: V920 | Cohort 1: Placebo | Cohort 2: V920 | Cohort 2: Placebo | Cohort 3: V920 | Cohort 3: Placebo | Cohort 4: V920 | Cohort 4: Placebo | Cohort 5: V920 | Cohort 5: Placebo | Total
Number analyzed (Participants) | 41 | 10 | 40 | 10 | 41 | 9 | 40 | 10 | 40 | 10 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 40 | 10 | 12 | 3 | 65
  Between 18 and 65 years | 40 | 10 | 39 | 10 | 41 | 9 | 0 | 0 | 28 | 7 | 184
  >=65 years | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (8.0) | 48.9 (8.6) | 48.1 (8.3) | 49.9 (7) | 46.6 (11.1) | 44.1 (8.8) | 15 (1.5) | 14.5 (1.4) | 33.1 (15.2) | 33.8 (19) | 44 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 6 | 24 | 7 | 18 | 6 | 20 | 7 | 21 | 4 | 130
  Male | 24 | 4 | 16 | 3 | 23 | 3 | 20 | 3 | 19 | 6 | 121
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 21 | 5 | 39 | 10 | 41 | 9 | 40 | 10 | 40 | 10 | 225
  Race: Multiple - Asian, White | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Race: White | 20 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 20 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26
  Burkina Faso | 12 | 3 | 23 | 6 | 25 | 6 | 38 | 9 | 24 | 6 | 152
  Senegal | 9 | 2 | 16 | 4 | 16 | 3 | 2 | 1 | 16 | 4 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events Following V920 Vaccination
Description: The number of participants with general solicited local (at the injection site) and systemic adverse events following vaccination will be summarized.
  Local AES include: pain at injection site, redness at injection site, swelling at injection site Systemic AEs include: fever, arthritis, arthralgia, rash and blisters/vesicular lesions.
Time Frame: From vaccine administration up to day 14 following vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  ≥500 cells/mm3 Adults.
- Cohort 2: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  >350 and <500 cells/mm3 Adults.
- Cohort 3: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  ≥200 and ≤350 cells/mm3 Adults.
- Cohort 4: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  ≥200 cells/mm3 Adolescents.
- Cohort 5: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  ≥200 cells/mm3 Adults and adolescents.
Arm/Group | Cohort 1: V920 | Cohort 1: Placebo | Cohort 2: V920 | Cohort 2: Placebo | Cohort 3: V920 | Cohort 3: Placebo | Cohort 4: V920 | Cohort 4: Placebo | Cohort 5: V920 | Cohort 5: Placebo
Number analyzed (Participants) | 40 | 10 | 40 | 10 | 41 | 9 | 40 | 10 | 40 | 10
Participants
  Local - injection site erythema | 5 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Local - Injection site pain | 22 | 3 | 20 | 3 | 24 | 1 | 34 | 3 | 30 | 2
  Local - Injection site swelling | 4 | 0 | 0 | 1 | 2 | 0 | 4 | 1 | 1 | 1
  Systemic - Abdominal pain | 4 | 0 | 5 | 1 | 4 | 1 | 4 | 1 | 8 | 1
  Systemic - Arthralgia | 14 | 0 | 16 | 2 | 7 | 1 | 3 | 0 | 10 | 1
  Systemic - Blister | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Systemic - Chills | 14 | 0 | 4 | 1 | 8 | 1 | 3 | 0 | 6 | 0
  Systemic - Diarrhea | 10 | 1 | 2 | 1 | 2 | 1 | 1 | 0 | 2 | 0
  Systemic - Fatigue | 21 | 3 | 18 | 5 | 24 | 1 | 8 | 1 | 20 | 1
  Systemic - Feeling hot | 11 | 0 | 7 | 2 | 8 | 1 | 10 | 3 | 15 | 1
  Systemic - Headache | 23 | 4 | 21 | 2 | 20 | 2 | 22 | 5 | 23 | 0
  Systemic - Hyperhidrosis | 11 | 0 | 1 | 0 | 3 | 1 | 4 | 0 | 7 | 1
  Systemic - Joint swelling | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Systemic - Myalgia | 12 | 2 | 8 | 1 | 2 | 0 | 3 | 0 | 10 | 0
  Systemic - Nausea | 10 | 1 | 3 | 2 | 3 | 0 | 3 | 0 | 9 | 0
  Systemic - Pyrexia | 5 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0
  Systemic - Rash | 1 | 1 | 2 | 2 | 1 | 1 | 2 | 1 | 2 | 0

2. Primary Outcome: Number of Participants With Solicited Adverse Events Following V920 Vaccination
Description: The number of participants with solicited systemic adverse events following vaccination that include arthralgia, blister, joint swelling, pyrexia and rash
Time Frame: From vaccine administration up to 42 days postvaccination
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  Adults CD4≥500
- Cohort 1: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adults CD4≥500
- Cohort 2: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  Adults CD4 >350 and <500
- Cohort 2: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adults CD4 >350 and <500
- Cohort 3: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  Adults CD4 ≥200 and ≤350
- Cohort 3: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adults CD4 ≥200 and ≤350
- Cohort 4: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  Adolescents CD4≥200
- Cohort 4: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adolescents CD4≥200
- Cohort 5: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine.
  Adults and Adolescents CD4≥200
- Cohort 5: Placebo: Participants randomly assigned to receive placebo.
  Saline: Normal saline (0.9%) was chosen as an inert substance to serve as placebo control.
  Adults and Adolescents CD4≥200
Arm/Group | Cohort 1: V920 | Cohort 1: Placebo | Cohort 2: V920 | Cohort 2: Placebo | Cohort 3: V920 | Cohort 3: Placebo | Cohort 4: V920 | Cohort 4: Placebo | Cohort 5: V920 | Cohort 5: Placebo
Number analyzed (Participants) | 40 | 10 | 40 | 10 | 41 | 9 | 40 | 10 | 40 | 10
Participants
  Arthralgia | 9 | 2 | 15 | 2 | 6 | 0 | 0 | 0 | 6 | 1
  Blister | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Joint swelling | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pyrexia | 8 | 0 | 2 | 0 | 1 | 0 | 7 | 0 | 3 | 0
  Rash | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 0

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events Following V920 Vaccination
Description: The number of participants with unsolicited adverse events following vaccination.
  These include the following disorders:
  Blood and lymphatic system disorders, cardiac disorders, ear and labyrinth disorders, eye disorders, gastrointestinal disorders, general disorders and administration site conditions, infections and infestations, injury, poisoning and procedural complications, metabolism and nutrition disorders, musculoskeletal and connective tissue disorders, nervous system disorders, psychiatric disorders, reproductive system and breast disorders, respiratory, thoracic and mediastinal disorders, skin and subcutaneous tissue disorders,vascular disorders.
Time Frame: From vaccine administration up to day 42 postvaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: V920 | Cohort 1: Placebo | Cohort 2: V920 | Cohort 2: Placebo | Cohort 3: V920 | Cohort 3: Placebo | Cohort 4: V920 | Cohort 4: Placebo | Cohort 5: V920 | Cohort 5: Placebo
Number analyzed (Participants) | 40 | 10 | 40 | 10 | 41 | 9 | 40 | 10 | 40 | 10
Participants
  Blood and lymphatic system disorders - Lymphadenopathy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac disorders - Angina pectoris | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Ear and labyrinth disorders - Cerumen impaction | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Eye disorders - Conjunctivitis allergic | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  Eye disorders - Eye irritation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Eye disorders - Eye pain | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Gastrointestinal disorders - Abdominal pain | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Gastrointestinal disorders - Abdominal pain upper | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Gastrointestinal disorders - Dental caries | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Gastrointestinal disorders - Diarrhea | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Gastrointestinal disorders - Dyspepsia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Gastroduodenal ulcer | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Gastrointestinal disorder | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Malpositioned teeth | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Oral papule | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Peptic ulcer | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Toothache | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  General disorders and administration site conditions - Chest pain | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  General disorders and administration site conditions - Fatigue | 6 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  General disorders and administration site conditions - Ill-defined disorder | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  General disorders and administration site conditions - Injection site induration | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  General disorders and administration site conditions - Pain | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  General disorders and administration site conditions - Tenderness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Amoebic dysentery | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Infections and infestations - Bronchitis | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 0
  Infections and infestations - Conjunctivitis | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0
  Infections and infestations - Conjunctivitis bacterial | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections and infestations - Cutaneous leishmaniasis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Infections and infestations - Cystitis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Furuncle | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Infections and infestations - Gastroenteritis | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Influenza | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Malaria | 5 | 1 | 1 | 0 | 1 | 0 | 4 | 1 | 2 | 0
  Infections and infestations - Nasopharyngitis | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Orchitis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Infections and infestations - Otitis media chronic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Infections and infestations - Parasitic gastroenteritis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Paronychia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Infections and infestations - Pilonidal disease | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Pneumonia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Rhinitis | 0 | 0 | 3 | 0 | 4 | 1 | 2 | 0 | 3 | 0
  Infections and infestations - Sinobronchitis | 0 | 0 | 1 | 0 | 4 | 1 | 3 | 0 | 1 | 0
  Infections and infestations - Tinea pedis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Tonsillitis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Tooth abscess | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Tooth infection | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Typhoid fever | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Upper respiratory tract infection | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Urinary tract infection | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Infections and infestations - Vulvovaginal mycotic infection | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications -Ankle fracture | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications - Limb injury | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
  Injury, poisoning and procedural complications - Thermal burn | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Metabolism and nutrition disorders - Decreased appetite | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders - Back pain | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders - Bursitis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders - Myalgia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders - Pain in extremity | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders - Torticollis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Nervous system disorders - Burning sensation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders - Carpal tunnel syndrome | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders - Dizziness | 0 | 0 | 4 | 0 | 3 | 0 | 1 | 0 | 0 | 1
  Nervous system disorders - Headache | 1 | 0 | 3 | 0 | 2 | 0 | 1 | 1 | 3 | 0
  Nervous system disorders - Cervicobrachial syndrome | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders - Intercostal neuralgia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders - Paraesthesia | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders - Sciatica | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Psychiatric disorders - Insomnia | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reproductive system and breast disorders - Breast pain | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reproductive system and breast disorders - Dysmenorrhoea | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Reproductive system and breast disorders - Heavy menstrual bleeding | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reproductive system and breast disorders - Vaginal discharge | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Bronchopneumopathy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Cough | 2 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 3 | 1
  Respiratory, thoracic and mediastinal disorders - Lung disorder | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Oropharyngeal pain | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Acne | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Ecchymosis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Hyperhidrosis | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Intertrigo | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Prurigo | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Pruritus | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
  Vascular disorders - Diastolic hypertension | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Vascular disorders - Hypertension | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Serious Adverse Events Following V920 Vaccination
Description: The number of participants with solicited vaccine-related serious adverse events following V920 vaccination.
Time Frame: From vaccine administration up to day 365 following vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: V920: Participants randomly assigned to receive ≥2 x 107 pfu of the V920 (rVSVΔG-ZEBOV-GP) Ebola Virus Vaccine
  ≥500 cells/mm3 Adults
Arm/Group | Cohort 1: V920 | Cohort 1: Placebo | Cohort 2: V920 | Cohort 2: Placebo | Cohort 3: V920 | Cohort 3: Placebo | Cohort 4: V920 | Cohort 4: Placebo | Cohort 5: V920 | Cohort 5: Placebo
Number analyzed (Participants) | 40 | 10 | 40 | 10 | 41 | 9 | 40 | 10 | 40 | 10
Participants | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

5. Primary Outcome: Geometric Mean Titers Induced by V920
Description: Geometric Mean Titers (GMTs) for ZEBOV-specific antibodies at Day 28 were calculated for each treatment group, along with two-sided 95% CIs, by exponentiating the corresponding log-transformed mean and two-sided 95% confidence limits.
  Cohorts 1-5.
Time Frame: Day 28 postvaccination
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 1: V920 | Cohort 1: Placebo | Cohort 2: V920 | Cohort 2: Placebo | Cohort 3: V920 | Cohort 3: Placebo | Cohort 4: V920 | Cohort 4: Placebo | Cohort 5: V920 | Cohort 5: Placebo
Number analyzed (Participants) | 40 | 10 | 40 | 10 | 41 | 9 | 40 | 10 | 40 | 10
Titer | 1655.0 [1,151.4 to 2,378.9] | 18.1 [8.7 to 37.3] | 1124.6 [821.0 to 1,540.4] | 26.8 [13.8 to 52.0] | 868.8 [679.0 to 1,111.6] | 29.7 [17.5 to 50.2] | 1432.8 [1,091.0 to 1,881.8] | 30.4 [17.6 to 52.4] | 1191.8 [865.7 to 1,640.6] | 43.1 [22.8 to 81.8]
Statistical Analysis 1: Comparison: Cohort 1: V920 vs Cohort 1: Placebo vs Cohort 2: V920 vs Cohort 2: Placebo vs Cohort 3: V920 vs Cohort 3: Placebo vs Cohort 4: V920 vs Cohort 4: Placebo vs Cohort 5: V920 vs Cohort 5: Placebo; V920 vs. placebo in Cohorts 1 to 5 combined; Test type: Superiority; p < 0.001, ANOVA; Fold difference = 42.90, 95% CI 2-sided [31.49 to 58.43]

6. Primary Outcome: Geometric Mean Titers Induced by V920
Description: Geometric Mean Titers (GMTs) for ZEBOV-specific antibodies at Day 28 were calculated for each treatment group, along with two-sided 95% CIs, by exponentiating the corresponding log-transformed mean and two-sided 95% confidence limits
  Only Cohort 5 received 2 doses of vaccine.
Time Frame: 28 days after LAST (second) dose of vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cohort 5: V920 | Cohort 5: Placebo
Number analyzed (Participants) | 40 | 10
Titer | 8,416.0 [6,461.9 to 10,961.1] | 40.3 [23.8 to 68.4]
Statistical Analysis 1: Comparison: Cohort 5: V920 vs Cohort 5: Placebo; Test type: Superiority; p < 0.001, ANOVA; Fold difference = 208.66, 95% CI 2-sided [115.57 to 376.72]

ADVERSE EVENTS:
Time Frame: 365 days
Description: Serious Adverse Events were monitored at every visit through Day 365.
  All-cause mortality reported are at 1-year post vaccination.
  SAEs reported in this section are at 1-year postvaccination.
  AEs reported in this section are at 42 days postvaccination.
Arm/Group | Cohort 1: V920 | Cohort 1: Placebo | Cohort 2: V920 | Cohort 2: Placebo | Cohort 3: V920 | Cohort 3: Placebo | Cohort 4: V920 | Cohort 4: Placebo | Cohort 5: V920 | Cohort 5: Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/10 | 0/40 | 0/10 | 0/41 | 0/9 | 0/40 | 0/10 | 0/40 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/10 | 0/40 | 0/10 | 1/41 | 0/9 | 0/40 | 1/10 | 0/40 | 0/10
Other Adverse Events (participants affected / at risk) | 25/40 | 5/10 | 11/40 | 4/10 | 8/41 | 5/9 | 20/40 | 4/10 | 13/40 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: V920 (N=40) | Cohort 1: Placebo (N=10) | Cohort 2: V920 (N=40) | Cohort 2: Placebo (N=10) | Cohort 3: V920 (N=41) | Cohort 3: Placebo (N=9) | Cohort 4: V920 (N=40) | Cohort 4: Placebo (N=10) | Cohort 5: V920 (N=40) | Cohort 5: Placebo (N=10)
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: V920 (N=40) | Cohort 1: Placebo (N=10) | Cohort 2: V920 (N=40) | Cohort 2: Placebo (N=10) | Cohort 3: V920 (N=41) | Cohort 3: Placebo (N=9) | Cohort 4: V920 (N=40) | Cohort 4: Placebo (N=10) | Cohort 5: V920 (N=40) | Cohort 5: Placebo (N=10)
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — 42 days post vaccination
Fatigue (General disorders) | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Malaria (Infections and infestations) | 5 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 0 — 42 days post vaccination
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 — 42 days post vaccination
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 3 | 1 — 42 days post vaccination
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 — 42 days post vaccination
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Pain (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 — 42 days post vaccination
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Dizziness (Nervous system disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — 42 days post vaccination
Headache (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 3 | 0 — 42 days post vaccination
Diastolic Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — 42 days post vaccination
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 0 | 3 | 0 — 42 days post vaccination
Sinobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 1 | 3 | 0 | 0 | 0 — 42 days post vaccination
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — 42 days post vaccination
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — 42 days post vaccination
Ill-defined Disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 — 42 days post vaccination
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — 42 days post vaccination
Otitis Medica Chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — 42 days post vaccination
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — 42 days post vaccination
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 — 42 days post vaccination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT03031912/Prot_SAP_001.pdf